CLINICAL TRIAL: NCT02215564
Title: Bordetella Pertussis Carriage in College-aged Students
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, J. Owen Hendley, MD, Professor of Pediatrics, University of Virginia
Other Study IDs: 17545
Record Dates: First submitted 2014-08-06; First posted 2014-08-13 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Carriage of Bordetella Pertussis
Keywords: Bordetella pertussis; Carriage rates in young adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: Young adults tested by PCR for B. pertussis carriage

SUMMARY:
The objective in this observational cohort study of young adults sampled at three intervals during the academic year is to ascertain if there is carriage of B. pertussis in asymptomatic individuals. We hypothesize that in asymptomatic college students there is no carriage of B. pertussis detectable by polymerase chain reaction (PCR) assay.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Not immunosuppressed
* Not HIV positive (not known to be/self-reported)
* Able to tolerate swab procedures
* Able to provide consent

Exclusion Criteria:

* No antimicrobial or immunosuppressive medications taken for chronic conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: College-aged students/young adults
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-06 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with B. pertussis by PCR in nasopharyngeal sample at first timepoint | 30 minutes
  Participants will be tested for B. pertussis by PCR at one visit in October 2014, 30 minutes.

SECONDARY OUTCOMES:
Number of participants with B. pertussis by PCR in nasopharyngeal sample at second timepoint | 30 minutes
  Participants will be tested for B. pertussis by PCR at one visit in January 2015, 30 minutes.

OTHER OUTCOMES:
Number of participants with B. pertussis by PCR in nasopharyngeal sample at third timepoint | 30 minutes
  Participants will be tested for B. pertussis by PCR at one visit in April 2015, 30 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Nuolivirta K, Koponen P, He Q, Halkosalo A, Korppi M, Vesikari T, Helminen M. Bordetella pertussis infection is common in nonvaccinated infants admitted for bronchiolitis. Pediatr Infect Dis J. 2010 Nov;29(11):1013-5. PMID 21046700
- [Background] Zhang Q, Yin Z, Li Y, Luo H, Shao Z, Gao Y, Xu L, Kan B, Lu S, Zhang Y, Li M, Liu M, Yao P, Zhao Z, He Q. Prevalence of asymptomatic Bordetella pertussis and Bordetella parapertussis infections among school children in China as determined by pooled real-time PCR: a cross-sectional study. Scand J Infect Dis. 2014 Apr;46(4):280-7. doi: 10.3109/00365548.2013.878034. Epub 2014 Feb 13. PMID 24520981